CLINICAL TRIAL: NCT03187639
Title: Fractional Flow Reserve Derived From Computed Tomography Coronary Angiography in the Assessment and Management of Stable Chest Pain
Acronym: FORECAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: The FORECAST Trial
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; CT coronary angiography; FFRct; Rapid access chest pain clinic; Stable chest pain; Resource utilisation; Quality of life
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: FORECAST is a randomised controlled trial comparing 1400 patients with new onset pain who are assigned to either routine assessment or FFRct assessment (n=700 per group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FFRct default primary investigation (Experimental): All patients undergo FFRct as the default test assuming they have no pre-specified contraindications to CT angiography. The result of the FFRct will be conveyed to the supervising physician within 24 hours and will be used to determine the subsequent management plan.
  Interventions: Diagnostic Test: FFRct
- Standard care (Active Comparator): All patients will be assessed and managed exactly as they are usually treated by the randomising centre and the RACP using the local algorithms interpreted from the NICE Chest Pain of Recent Onset Guidance.
  Interventions: Diagnostic Test: Standard care

INTERVENTIONS:
Diagnostic Test: FFRct — In the test group all patients who are eligible for CTA will undergo CTA as their default test. Those patients with any coronary stenosis of equal or > 40% data in at least one major epicardial vessel of stentable/graftable diameter will be referred for FFRct. (NB Lesions in distal vessels or vessels of a diameter not suitable for stenting/grafting will not qualify for FFRct if there are no other more significant lesions). In patients in whom FFRct analysis is performed, FFR will be derived for all vessels. The data derived from this test will determine their management strategy. The patients in this arm will not follow the NICE guideline algorithm. Those patients randomised to FFRct with contraindications for CTA will be asked to take part in a trial registry.
  Arms: FFRct default primary investigation
Diagnostic Test: Standard care — All patients in the standard care group will be assessed according to their current conventional pathways that are based upon NICE guidelines for Chest Pain of Recent Onset. The trial will encourage the routine and standard assessment and management of all patients at these sites… (anticipated outcomes include ETT, stress echo, stress MR, nuclear perfusion, CTA, CT calcium, invasive CA, reassurance), in accordance with the local application of the NICE guideline for chest pain of recent onset.
  Arms: Standard care

SUMMARY:
To determine whether, in a population of patients presenting to the rapid access chest pain clinic (RACPC), routine FFRct (Fractional Flow Reserve Computed Tomography) as a default test is superior in terms of resource utilisation when compared to routine clinical pathway algorithms recommended by the National Institute for Health and Care Excellence (NICE)

DETAILED DESCRIPTION:
FORECAST is a randomised controlled trial comparing 1400 patients with new onset pain who are assigned to either routine assessment or FFRct assessment.

This trial aims to test the hypothesis that FFRct, used as the default screening tool for patients presenting with new onset stable chest pain, would be associated with (i) shorter time period between initial consultation and definitive management plan; (ii) better patient experience; (iii) lower overall use of resources.

The UK is well suited to test this hypothesis because of its well established system of Rapid Access Chest Pain Clinics (RACPC). The majority of patients presenting with stable chest pain (CP) that is of suspected cardiac origin are referred to such clinics, with a mandated access time within 2 weeks. The majority of such clinics work to the algorithm recommended in the NICE guidelines for Chest Pain of Recent Onset (March 2010). Within this guideline, patients are stratified according to their risk profile and pre-test likelihood of coronary artery disease (CAD) to outcomes that include discharge, stress test, CTCA (computed tomography coronary angiography), CT (computed tomography) coronary calcium score and invasive coronary angiogram.

Given the relative streamlining of this initial assessment of such patients throughout the country, it facilitates a comparison of strategies in FORECAST.

Once eligibility for the trial is confirmed and informed consent received, patients will be enrolled in the study and randomised to a treatment group (1:1 ratio)

The 2 strategies for the FORECAST trial are:

[A] TEST: all patients undergo FFRct as the default test, assuming they have no prespecified contraindications to CT coronary angiography. The result of the FFRct will be conveyed to the supervising physician within 24 hours and will be used to determine the subsequent management plan.

[B] REFERENCE: all patients will be assessed and managed exactly as they are usually treated by that centre and that RACP using the local algorithms interpreted from the NICE Chest Pain of Recent Onset Guidance.

All patients in the "routine" assessment group (group B) will be assessed according to their current conventional pathways that are based upon NICE guidelines for Chest Pain of Recent Onset. The trial will encourage the routine and standard assessment and management of all patients at these site, (anticipated outcomes include exercise tolerance testing (ETT), stress echo, stress magnetic resonance imaging (MR), nuclear perfusion, CTA, CT calcium score, invasive coronary angiography, reassurance), in accordance to the local application of the NICE guideline for chest pain of recent onset.

In the FFRct group, all patients who are eligible for CTA will undergo CTA as their default test. Those patients with any coronary stenosis of equal to or >40% data in at least one major epicardial vessel of stentable/graftable diameter will be referred for FFRct. (NB Lesions in distal vessels or vessels of a diameter not suitable for stenting/grafting will not qualify for FFRct if there are no other more significant lesions). In patients in whom FFRct analysis is performed, FFR will be derived for all vessels. The data derived from this test will determine their management strategy. The patients in this arm will not follow the NICE guideline algorithm. Those patients randomised to FFRct with contraindications for CTA will be asked to take part in a trial registry.

Data will be collected according to detailed specialised methodology for tracking of (i) resource utilisation including all cardiac-related medications, tests, hospital visits; (ii) QOL; (iii) clinical events as described above.

Data collection will occur at 3 and 9 month timepoints

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18
* Primary symptom of chest pain
* No contraindication to CTA
* Willing and able to provide written informed consent

Exclusion Criteria:

* Atrial fibrillation of new onset or when rate control has been difficult
* Known bigemini/trigeminy
* Prior CABG surgery
* Allergic to contrast
* Advanced renal impairment
* Significant valve disease (severe aortic stenosis or regurgitation; severe mitral regurgitation)
* Life expectancy <12 months
* Inclusion in another trial without prior agreement with CI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Resource utilisation | 9 months
  To determine whether, in a population of patients presenting to RACPC, routine FFRct as a default test is superior, in terms of resource utilisation, when compared to routine clinical pathway algorithms recommended by NICE.

SECONDARY OUTCOMES:
Quality of Life | 9 months
  Seattle angina questionnaire, EQ-5D, illness perception
MACE | 9 months
  Myocardial infarction, all cause death, unplanned coronary revascularisation

CONTACTS AND LOCATIONS:
Locations (1):
- Southampton Clinical Trials Unit, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hlatky MA, Wilding S, Stuart B, Nicholas Z, Shambrook J, Eminton Z, Fox K, Connolly D, O'Kane P, Hobson A, Chauhan A, Uren N, Mccann GP, Berry C, Carter J, Roobottom C, Mamas M, Rajani R, Ford I, Douglas PS, Curzen N. Randomized comparison of chest pain evaluation with FFRCT or standard care: Factors determining US costs. J Cardiovasc Comput Tomogr. 2023 Jan-Feb;17(1):52-59. doi: 10.1016/j.jcct.2022.09.005. Epub 2022 Sep 24. PMID 36216700